CLINICAL TRIAL: NCT06239974
Title: Randomised Controlled Trial of Vericiguat in Patients With Coronary Microvascular Dysfunction Causing Stable Chest Pain (V-COM)
Brief Title: Vericiguat in Patients With Coronary Microvascular Dysfunction Causing Stable Chest Pain (V-COM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: UW 23-605
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2024-11

CONDITIONS: Chest Pain
Keywords: Stress Cardiac Magnetic Resonance
MeSH Terms: conditions — Chest Pain | interventions — vericiguat

STUDY DESIGN:
Intervention Model Description: Single-blinded Randomised Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Cardiovascular Magnetic Resonance Level 3 radiologists will be blinded to the patient allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Patients will have no intervention and will continue to have optimised medical therapy and follow-up appointments (currently 1 appointment every 3 months).
  Interventions: Diagnostic Test: Stress Cardiac Magnetic Resonance
- Intervention group (Experimental): Patients will be prescribed vericiguat once a day for 6 months, starting at 2.5mg and titrated up to the full dose of 10mg per day (doubling of dose every 2 weeks) in addition to optimised medical therapy and standard follow-up like the control group
  Interventions: Drug: Vericiguat; Diagnostic Test: Stress Cardiac Magnetic Resonance

INTERVENTIONS:
Drug: Vericiguat — Patients will be prescribed vericiguat once a day for 6 months, starting at 2.5mg and titrated up to the full dose of 10mg per day (doubling of dose every 2 weeks) in addition to optimised medical therapy and standard follow-up like the control group
  Other Names: Verquvo
  Arms: Intervention group
Diagnostic Test: Stress Cardiac Magnetic Resonance — All patients will have stress CMR examinations at recruitment and at the end of trial.
  Other Names: Stress CMR

SUMMARY:
This is a randomised controlled trial to determine the effectiveness of Vericiguat to improve stress myocardial blood flow (MBF) and myocardial perfusion reserve as measured by cardiac magnetic resonance (CMR) imaging.

DETAILED DESCRIPTION:
Stable chest pain is one of the most common complaints by patients. However, about 50% of patients referred for catheter coronary angiograms do not have obstructive coronary artery disease (CAD). In the United Kingdom (UK), one very large population study showed that ~70% of patients did not have a cause for the chest pain diagnosed within 6 months of presentation. Furthermore, the study further showed that this group of patients had a significantly higher risk of major adverse cardiovascular events (MACE) compared to patients without chest pain. It is now understood that the two major causes of cardiac chest pain with non obstructive CAD (also known as Ischaemia with Non Obstructive Coronary Arteries (INOCA)) are coronary microvascular dysfunction (CMD) and the other is coronary vasospasm. CMD and coronary vasospasm have been shown in one randomised controlled study to comprise 52% and 17% of all patients with INOCA. However, therapies for CMD are lacking and has been highlighted as a major area of need.

ELIGIBILITY:
Inclusion Criteria:

1. Stable recurrent chest pain.
2. 40 to 75 years old.
3. Have coronary computed tomography (CT) angiogram or catheter coronary angiogram within 6 months showing non-obstructive coronary artery disease (<50% coronary artery stenosis or fractional flow reserve >0.8).
4. Stress CMR MPR <2.19 12 or Stress MBF <2.19ml/g/min 13.
5. Female participant is eligible to participate if she is not pregnant or breastfeeding, is not a woman of childbearing potential (WOCBP),or is a WOCBP and agrees to follow contraceptive guidance during the study intervention period and for at least 1 month after the last dose of study intervention.

Exclusion Criteria:

1. Systolic blood pressure <100 mm Hg.
2. Concurrent use of soluble guanylate cyclase stimulators (eg. Riociguat), or phosphodiesterase type 5 inhibitors (eg. vardenafil, tadalafil, and sildenafil).
3. Has known allergy or sensitivity to any soluble guanylate cyclase stimulator.
4. On long-acting nitrates (eg. isosorbide mononitrate)
5. Known cardiomyopathy, complex congenital heart disease, endocarditis or pericarditis.
6. Has acute coronary syndrome (unstable angina, non-ST elevation myocardial infarction (NSTEMI), or ST elevation myocardial infarction (STEMI)) or coronary revascularization (coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI)) within 60 days prior to randomisation, or indication for coronary revascularization at time of randomisation.
7. Has symptomatic carotid stenosis, transient ischemic attack (TIA) or stroke within 60 days prior to randomisation.
8. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2
9. Malignancy or other non-cardiac condition limiting life expectancy to <3 years.
10. Patient's with implanted devices which are not MRI compatible.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Difference in stress myocardial blood flow (MBF) | 36 months
  Difference in stress MBF as measured by stress CMR between patients receiving Vericiguat and patients not receiving Vericiguat
Difference in stress myocardial perfusion reserve (MPR) | 36 months
  Difference in stress MPR as measured by stress CMR between patients receiving Vericiguat and patients not receiving Vericiguat

SECONDARY OUTCOMES:
Improvement in exercise tolerance through performing a cardiopulmonary exercise test. | 36 months
  Measured by baseline and end of study 6-minute walk test
Progression in patient symptoms diagnoses. | 36 months
  The Seattle Angina Questionnaire (SAQ-7) scores are transformed to a range of 0-100, in which higher scores reflect better health status. The measurement will take place at time of baseline CMR and at follow-up CMR in order to determine if there is an improvement in patient symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No